CLINICAL TRIAL: NCT04759625
Title: Development of a Novel Biscuit Enriched With β-glucans Isolated From Edible Mushrooms of Greek Habitats and Implementation of a Dietary Intervention That Includes Daily Consumption of This Biscuit
Brief Title: Effect of Daily Consumption of a Novel Biscuit Enriched With Edible Mushrooms, on Intestinal Health-related Parameters
Acronym: FUNglucan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: Agricultural University of Athens (Other); National Hellenic Research Foundation (Other); PAPADOPOULOS S.A (Unknown)
Responsible Party: Principal Investigator, Adamantini Kyriakou, Associate Professor, Harokopio University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: T1EDK-03404
Record Dates: First submitted 2021-02-03; First posted 2021-02-18 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: β-glucans; edible mushrooms; functional food; prebiotic activity; gut microbiota; older adults

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biscuit enriched with mushroom powder (Experimental): Daily consumption of a novel biscuit enriched with mushroom powder containing 3g of β-glucans
  Interventions: Other: Novel biscuit enriched with mushroom powder containing 3g of β-glucans
- Placebo biscuit (Placebo Comparator): Daily consumption of a placebo biscuit
  Interventions: Other: Placebo biscuit

INTERVENTIONS:
Other: Novel biscuit enriched with mushroom powder containing 3g of β-glucans — Daily consumption of a novel biscuit enriched with mushroom powder containing 3g of β-glucans
  Arms: Biscuit enriched with mushroom powder
Other: Placebo biscuit — Daily consumption of placebo biscuit
  Arms: Placebo biscuit

SUMMARY:
The purpose of the study is to assess the effect of dietary intervention that includes the daily consumption of a novel biscuit (enriched with the selected mushrooms rich in β-glucans) on gut health related parameters of healthy subjects over 60 years old.

DETAILED DESCRIPTION:
After having been informed about the study and the potential risks, all subjects giving written informed consent will undergo screening to determine eligibility for study entry (inclusion criteria). At baseline, the participants will provide biological samples and they will be randomly assigned in a double-blind manner (investigator and participant) to one of the intervention groups, i.e. consumption of the novel biscuit (biscuit enriched with mushroom powder containing 3g of β-glucans) or consumption of the placebo biscuit for 3 months,. After a washout period of 2 months, the subjects will consume the novel biscuit or the placebo biscuit in a cross-over design for 3 more months. Throughout the interventional period subjects' dietary intake, anthropometrical data and gastrointestinal symptoms will be monitored. Meanwhile at baseline and at the end of each trimester physical activity, mental health and sleep habits will be evaluated with the use of questionnaires and biological samples will be provided for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals aged 60-80 years old, of both sexes/genders

Exclusion Criteria:

* no recent weight loss and extreme dietary behaviors;
* no history of gastrointestinal disease, chronic constipation, chronic/acute diarrhea, autoimmune disease, coronary disease, liver and/or kidney malfunction;
* no consumption of antibiotics two months prior to the initiation of the intervention;
* no consumption of probiotics and/or prebiotics and/or dietary fiber supplements two weeks prior to the initiation of the intervention.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Gastrointestinal tolerance of novel biscuit during the interventional period and at 3 months. | Gastrointestinal symptoms will be evaluated at baseline, during and at the end of each intervention. (3 months period)
  Gastrointestinal (GI) symptomatology will be recorded through a 7d-questionnaire in certain time periods.The intensity of each GI symptom (abdominal pain, distension, ﬂatulence and borborygmi) will be measured daily on a scale of 0-4, where '0' represents absence of symptoms and '4' severe symptoms. The possible range for each weekly symptom score is 0-28, and for the total symptom score 0-112. Frequency and consistency of evacuations will be also noted, and presence of diarrhoea will be defined.
Change from baseline to the effect on the intestinal microbial populations and their metabolic products [i.e. Short-Chain Fatty Acids (SCFA)] (prebiotic effect) at 3 months. | The levels of microbial populations and their metabolic products e.g. SCFA will be measured at baseline and at the end of each interventional period.(3 months period)
  Microbial populations will be quantified with 16SRNA sequencing and quantitative Polymerase Chain Reaction (PCR). SCFAs will be quantified with Gas chromatography.

SECONDARY OUTCOMES:
Change from baseline in Metabolic health at 3 months. | Metabolic health will be measured at baseline and at the end of each interventional period.(3 months period)
  Blood samples will be obtained after an overnight, 12-h fasting. Blood serum analysis will include assessment of lipidemic profile [i.e. Total Cholesterol (TC), Low-Density Lipoprotein Cholesterol (LDL-C), High-Density Lipoprotein Cholesterol (HDL-C), Triglycerides (TG)], glucose metabolism [i.e. Fasting Blood Glucose (FBG)] and uric acid. (units of measure: mg/dL)
Change from baseline in blood serum Insulin at 3 months. | Blood serum Insulin will be measured at baseline and at the end of each interventional period.(3 months period)
  Blood samples will be obtained after an overnight, 12-h fasting. Blood serum analysis will include assessment of glucose metabolism [i.e. Insulin (INS)]. (units of measure: μIU/mL)
Change from baseline in blood serum 25-hydroxy vitamin D at 3 months. | Blood serum 25-hydroxy vitamin D will be measured at baseline and at the end of each interventional period.(3 months period)
  Blood samples will be obtained after an overnight, 12-h fasting. Blood serum analysis will include assessment of bone biomarkers (i.e. 25-hydroxy vitamin D).(units of measure: ng/mL)
Change from baseline in blood serum Parathyroid Hormone at 3 months. | Blood serum Parathyroid Hormone will be measured at baseline and at the end of each interventional period.(3 months period)
  Blood samples will be obtained after an overnight, 12-h fasting. Blood serum analysis will include assessment of bone biomarker [i.e. Parathyroid Hormone (PTH)].(units of measure: pg/mL)
Change from baseline in Immune system reinforcement at 3 months. | Immune system reinforcement will be measured at baseline and at the end of each interventional period.(3 months period)
  The production of Interleukins (IL) (i.e. IL-1β, IL-6, IL-10) and Tumor-necrosis factor alpha (TNF-a) in vitro by peripheral blood mononuclear cells (PBMCs) cultured and isolated from healthy immunocompetent subjects, after mitogen stimulation, will be determined in cell culture supernatants by ELISA techniques with commercially available kits. The cytokine expression levels will be determined in cell pellets by Quantitative Real Time Polymerase Chain Reaction (qRT-PCR). Concomitantly, the levels of the same cytokines will be assessed by ELISA in the serum collected from the same subjects.
Change from baseline in Dietary intake at 3 months. | Dietary intake will be measured at baseline and at the end of each interventional period.(3 months period)
  Dietary intake will be evaluated with the use of 3-days (2-weekdays and 1 weekend day) diet intake records.

CONTACTS AND LOCATIONS:
Overall Officials: Adamantini Kyriacou, Principal Investigator — Harokopio University of Athens
Locations (1):
- Harokopio University, Kallithea, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitsou EK, Saxami G, Stamoulou E, Kerezoudi E, Terzi E, Koutrotsios G, Bekiaris G, Zervakis GI, Mountzouris KC, Pletsa V, Kyriacou A. Effects of Rich in Beta-Glucans Edible Mushrooms on Aging Gut Microbiota Characteristics: An In Vitro Study. Molecules. 2020 Jun 18;25(12):2806. doi: 10.3390/molecules25122806. PMID 32570735
- [Background] Boulaka A, Christodoulou P, Vlassopoulou M, Koutrotsios G, Bekiaris G, Zervakis GI, Mitsou EK, Saxami G, Kyriacou A, Zervou M, Georgiadis P, Pletsa V. Genoprotective Properties and Metabolites of beta-Glucan-Rich Edible Mushrooms Following Their In Vitro Fermentation by Human Faecal Microbiota. Molecules. 2020 Aug 4;25(15):3554. doi: 10.3390/molecules25153554. PMID 32759726
- [Background] Mitsou EK, Kakali A, Antonopoulou S, Mountzouris KC, Yannakoulia M, Panagiotakos DB, Kyriacou A. Adherence to the Mediterranean diet is associated with the gut microbiota pattern and gastrointestinal characteristics in an adult population. Br J Nutr. 2017 Jun;117(12):1645-1655. doi: 10.1017/S0007114517001593. PMID 28789729
- See also: Project's official website. — https://funglucan.hua.gr/
- See also: Project's official facebook website. — https://www.facebook.com/FUNglucan-2604410072963486/
- See also: Project's official instagram website. — https://www.instagram.com/funglucan/

DOCUMENTS (3):
  • Study Protocol (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT04759625/Prot_002.pdf
  • Statistical Analysis Plan (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT04759625/SAP_003.pdf
  • Informed Consent Form (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT04759625/ICF_004.pdf